CLINICAL TRIAL: NCT07007637
Title: A Phase 3, Multicenter, Open-label Extension Study to Evaluate the Long-term Safety, Tolerability, and Efficacy of Subcutaneous Sonelokimab in Participants With Moderate to Severe Hidradenitis Suppurativa
Brief Title: A Study to Evaluate the Long-term Safety, Tolerability, and Efficacy of Subcutaneous Sonelokimab in Participants With Moderate to Severe Hidradenitis Suppurativa
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: MoonLake Immunotherapeutics AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M1095-HS-303; VELA-OLE (Other: Sponsor)
Record Dates: First submitted 2025-05-28; First posted 2025-06-06 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Hidradenitis Suppurativa
Keywords: Hidradenitis Suppurativa; Hidradenitis; Sweat Gland Diseases; Skin Diseases; Skin Diseases, Bacterial; Suppuration; Anti-Inflammatory Agents; Sonelokimab; Nanobody; Apocrine Gland Disease
MeSH Terms: conditions — Hidradenitis Suppurativa; Hidradenitis; Sweat Gland Diseases; Skin Diseases; Skin Diseases, Bacterial; Suppuration | interventions — sonelokimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: sonelokimab (Experimental): All participants will receive sonelokimab 120 mg Q4W for up to 2 years
  Interventions: Drug: Sonelokimab

INTERVENTIONS:
Drug: Sonelokimab — Sonelokimab

SUMMARY:
This is a study to evaluate the long-term safety, tolerability, and efficacy of sonelokimab in participants with moderate to severe hidradenitis suppurativa who were previously enrolled in a parental study.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have completed a parental study (M1095-HS-301 or M1095-HS-302 [adult studies] or M1095-HS-304 [adolescent study]) and are eligible to continue to receive sonelokimab at the time of completing the parental study.
* Female participants are eligible to participate if they are not pregnant or breastfeeding
* Male participants must be willing to use a condom when sexually active with a partner of childbearing potential . Male participants must also agree to refrain from donating sperm during the study and for at least 8 weeks after the last dose of study treatment.

Exclusion Criteria:

* Participants who meet any of the discontinuation criteria of the parental study at the time of enrollment in this OLE study.
* Participants who have ongoing or planned to use one or more of the prohibited HS or non-HS treatments specified in the protocol.
* Participants who plan to participate in another interventional study for a drug or device during this study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 835 (Estimated)
Dates: Start 2025-06-27 (Actual); Primary Completion 2028-06-13 (Estimated); Study Completion 2028-06-13 (Estimated)

PRIMARY OUTCOMES:
Long-term safety and tolerability of sonelokimab: Adverse events (AEs) following treatment with sonelokimab | 2.5-3 years
  Incidence, relatedness, severity and seriousness of all AEs
Long-term safety and tolerability of sonelokimab: Treatment emergent adverse events (TEAEs) | 2.5-3 years
  Incidence, relatedness, severity and seriousness of all TEAEs
Long-term safety and tolerability of sonelokimab: Adverse events of special interest (AESIs) | 2.5-3 years
  Incidence, relatedness, severity and seriousness of all AESIs
Long-term safety and tolerability of sonelokimab: Discontinuation of sonelokimab treatment due to AEs | 2.5-3 years
  Number of participants discontinued from sonelokimab treatment due to AEs
Long-term safety and tolerability of sonelokimab: Clinically significant changes in clinical laboratory parameters | 2.5-3 years
  Number of participants with clinically significant changes in hematology, biochemistry and urinalysis from baseline
Long-term safety and tolerability of sonelokimab: Clinically significant changes in vital signs and standard 12-lead electrocardiogram | 2.5-3 years
  Number of participants with clinically significant changes in vital signs and 12-lead ECG intervals from baseline

SECONDARY OUTCOMES:
Long-term efficacy of sonelokimab: Hidradenitis Suppurativa Clinical Response 75 (HiSCR75) | 2.5 - 3 years
  Percentage of participants achieving a HiSCR75 response over time
Long-term efficacy of sonelokimab: Hidradenitis Suppurativa Clinical Response 90 (HiSCR90) and 50 (HiSCR50) | 2.5 - 3 years
  Percentage of participants achieving a HiSCR90 and HiSCAR50 response over time
Long-term efficacy of sonelokimab: International Hidradenitis Suppurativa Severity Score System (IHS4) | 2.5 - 3 years
  Absolute change in IHS4 score over time
Long-term efficacy of sonelokimab: Number of abscesses, draining fistulas/tunnels; inflammatory nodules | 2.5 - 3 years
  Absolute change in number of abscesses, draining fistulas/tunnels; inflammatory nodules
Long-term efficacy of sonelokimab: Dermatology Life Quality Index (DLQI) | 2.5 - 3 years
  Change in DLQI total score
Long-term efficacy of sonelokimab: Hidradenitis Suppurativa Quality of Life (HiSQOL) | 2.5 - 3 years
  Change in HiSQOL total score

CONTACTS AND LOCATIONS:
Locations (23):
- United States (16):
  - Clinical Site, Birmingham, Alabama
  - Clinical Site, Northridge, California
  - Clinical Site, North Miami Beach, Florida
  - Clinical Site, Macon, Georgia
  - Clinical Site, Sandy Springs, Georgia
  - Clinical Site, Columbus, Indiana
  - Clinical Site, New Albany, Indiana
  - Clinical Site, Murray, Kentucky
  - Clinical Site, Canton, Michigan
  - Clinical Site, Clarkston, Michigan
  - Clinical Site, Waterford, Michigan
  - Clinical Site, New Brighton, Minnesota
  - Clinical Site, Omaha, Nebraska
  - Clinical Site, Murfreesboro, Tennessee
  - Clinical Site, Dallas, Texas
  - Clinical Site, San Antonio, Texas
- Canada (7):
  - Clinical Site, Fredericton, New Brunswick
  - Clinical Site, Barrie, Ontario
  - Clinical Site, Guelph, Ontario
  - Clinical Site, Markham, Ontario
  - Clinical Site, Peterborough, Ontario
  - Clinical Site, Toronto, Ontario
  - Clinical Site, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No